CLINICAL TRIAL: NCT05376449
Title: The Effect of an Adaptive Exercise Program on Chronic Inflammation in Spinal Cord Injury
Brief Title: Spinal Cord Injury - Exercise
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: HealthPartners Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A21-009
Record Dates: First submitted 2022-05-11; First posted 2022-05-17 (Actual); Results first posted 2025-10-20 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-09

CONDITIONS: Spinal Cord Injuries
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate start (Experimental): Intervention to start immediately after first visits.
  Interventions: Behavioral: HealthPartners NeuroWell Exercise Program
- Delayed start (Active Comparator): Intervention to start after 12 weeks delay.
  Interventions: Behavioral: HealthPartners NeuroWell Exercise Program

INTERVENTIONS:
Behavioral: HealthPartners NeuroWell Exercise Program — A 12-week exercise program geared towards individuals with neurological disorders or injuries run by the Regions Hospital Rehabilitation department at the HealthPartners Neuroscience Center. The exercise programming will be designed by the exercise physiologists and adapted to individuals' abilities. Exercise prescriptions will be designed based on established guidelines, level and completeness of injury, individual functional ability, individual goals, and baseline exercise assessments. Program will consist of strength and endurance adaptive exercise.

SUMMARY:
Long lasting inflammation in the body is related to cardiovascular and respiratory disease, which are the two most common causes of death in people living with spinal cord injury (SCI). Individuals with SCI have been reported to have higher levels of inflammation when compared to healthy individuals. Exercise is a well-known method to reduce inflammation; however, people with SCI are often inactive. The main goal of this study is to determine whether a 12-week adaptive exercise program can reduce inflammation in people with SCI. Participants will be randomized to start exercise immediately or after a 12-week delay.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide and provision of signed and dated informed consent form
* Age 18-70
* Diagnosis of SCI and post injury ≥ 6 months
* Able to achieve adequate active range of motion at the elbow and wrist (flexion/extension) and able to achieve at least 90° active shoulder flexion, in order to complete study activities

Exclusion Criteria:

* Non-English speaking
* Exercise program participation ≤1 month from study enrollment or any other exercise participation during the duration of the study
* Patients with significant cognitive impairment of any etiology that prevents them from being able to participate
* Patients that were given sternal or spinal precautions that would prevent excessive twisting, bending, overhead reaching and lifting over 10 pounds
* Patients with a history heart failure, chronic lung disease, angina or any other condition that causes unreasonable shortness of breath on exertion
* Has been diagnosed with autonomic dysreflexia that is severe, unstable, and uncontrolled
* Requires ventilator support
* Spasms that limit the ability of the subjects to participate in the study training as determined by the Investigator
* Pregnant, planning to become pregnant
* Any other medical conditions that could affect their ability to participate in the exercise program (as determined by study investigators)
* Active participation or past participation ≤3 months in any other interventional study.
* Unwilling to participate in all study related activities

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2022-05-09 (Actual); Primary Completion 2024-06-20 (Actual); Study Completion 2024-09-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amanda A Herrmann, PhD, Principal Investigator — HealthPartners Neuroscience Research
Locations (1):
- HealthPartners Neuroscience Center, Saint Paul, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Weeks 1-12
Arm/Group | Immediate Start | Delayed Start
Started | 12 | 12
Completed | 9 | 8
Not Completed | 3 | 4
Period: Weeks 13-24
Arm/Group | Immediate Start | Delayed Start
Started | 9 | 8
Completed | 9 | 5
Not Completed | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Immediate Start | Delayed Start | Total
Number analyzed (Participants) | 12 | 12 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 57 (11) | 49 (14) | 53 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 5 | 7
  Male | 10 | 7 | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 12 | 12 | 24
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race (NIH/OMB): American Indian or Alaska Native | 0 | 0 | 0
  Race (NIH/OMB): Asian | 0 | 1 | 1
  Race (NIH/OMB): Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Race (NIH/OMB): Black or African American | 2 | 1 | 3
  Race (NIH/OMB): White | 10 | 9 | 19
  Race (NIH/OMB): Some Other Race | 0 | 1 | 1
American Spinal Injury Association (ASIA) [Count of Participants; unit: Participants] — ASIA Impairment Scale A - Complete Injury B - Sensory Incomplete C - Motor Incomplete (Limited Movement) D - Motor Incomplete (Functional Movement) E - Normal Function
  Participants
    A | 1 | 5 | 6
    B | 0 | 0 | 0
    C | 4 | 2 | 6
    D | 4 | 3 | 7
    E | 0 | 0 | 0
    Unknown | 3 | 2 | 5
Neurological Level of Injury [Count of Participants; unit: Participants] — Neurological injury level describes the specific location where the spinal cord is damaged.
  C1-C8: Cervical T1-T12: Thoracic L1-L5: Lumbar S1-S5: Sacrum
  Participants
    C1-C8 | 10 | 3 | 13
    T1-T12 | 1 | 8 | 9
    L1-L5 | 0 | 0 | 0
    S1-S5 | 0 | 0 | 0
    Unknown | 1 | 1 | 2
Time Since Injury [Mean (Standard Deviation); unit: months] | 7 (8) | 13 (15) | 10 (12)
Ambulation [Count of Participants; unit: Participants]
  Ambulatory & Manual Wheelchair | 3 | 1 | 4
  Ambulatory Only | 3 | 3 | 6
  Ambulatory, Manual, and Power Wheelchairs | 2 | 0 | 2
  Manual and Power Wheelchairs | 2 | 4 | 6
  Manual Wheelchair Only | 0 | 3 | 3
  Power Wheelchair Only | 2 | 1 | 3
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg per square meter] | 27 (5) | 29 (7) | 28 (6)

OUTCOME MEASURES:

1. Primary Outcome: Effect of Exercise on Inflammation (C-reactive Protein)
Description: Change in C-reactive protein after 12 week exercise program
Time Frame: 12 weeks
Measure: Mean (Inter-Quartile Range); unit: mg/dL
Arm/Group | Immediate Start | Delayed Start
Number analyzed (Participants) | 9 | 8
mg/dL | 0.00 [-0.010 to 0.010] | 0.05 [0.00 to 0.55]

2. Primary Outcome: Effect of Exercise on Inflammation (Interleukin 6)
Description: Change in Interleukin 6 after 12 week exercise program
Time Frame: 12 weeks
Measure: Mean (Inter-Quartile Range); unit: pg/mL
Arm/Group | Immediate Start | Delayed Start
Number analyzed (Participants) | 8 | 8
pg/mL | -0.33 [-1.28 to -0.18] | 0.50 [0.03 to 1.84]

3. Primary Outcome: Effect of Exercise on Inflammation (Tumor Necrosis)
Description: Change in Tumor Necrosis Biomarker after 12 week exercise program
Time Frame: 12 weeks
Measure: Mean (Inter-Quartile Range); unit: pg/mL
Arm/Group | Immediate Start | Delayed Start
Number analyzed (Participants) | 8 | 8
pg/mL | -2 [-3 to 6] | 2 [-2 to 5]

ADVERSE EVENTS:
Time Frame: 24 weeks
Groups:
- Immediate Start - Exercise Program: Intervention to start immediately after first visits.
  HealthPartners NeuroWell Exercise Program: A 12-week exercise program geared towards individuals with neurological disorders or injuries run by the Regions Hospital Rehabilitation department at the HealthPartners Neuroscience Center. The exercise programming will be designed by the exercise physiologists and adapted to individuals' abilities. Exercise prescriptions will be designed based on established guidelines, level and completeness of injury, individual functional ability, individual goals, and baseline exercise assessments. Program will consist of strength and endurance adaptive exercise.
- Immediate Start - No Exercise: Intervention to start immediately after first visits - Delay after program is complete.
- Delayed Start - No Exercise: Intervention to start after 12 weeks delay.
- Delayed Start - Exercise Program: Intervention to start after 12 weeks delay.
  HealthPartners NeuroWell Exercise Program: A 12-week exercise program geared towards individuals with neurological disorders or injuries run by the Regions Hospital Rehabilitation department at the HealthPartners Neuroscience Center. The exercise programming will be designed by the exercise physiologists and adapted to individuals' abilities. Exercise prescriptions will be designed based on established guidelines, level and completeness of injury, individual functional ability, individual goals, and baseline exercise assessments. Program will consist of strength and endurance adaptive exercise.
Arm/Group | Immediate Start - Exercise Program | Immediate Start - No Exercise | Delayed Start - No Exercise | Delayed Start - Exercise Program
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/9 | 0/12 | 0/8
Serious Adverse Events (participants affected / at risk) | 2/12 | 0/9 | 3/12 | 2/8
Other Adverse Events (participants affected / at risk) | 9/12 | 2/9 | 4/12 | 5/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Immediate Start - Exercise Program (N=12) | Immediate Start - No Exercise (N=9) | Delayed Start - No Exercise (N=12) | Delayed Start - Exercise Program (N=8)
Acute intracranial hemorrage (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin Issues (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Infection around pacemaker
Lighheaded/Syncope (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infection (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Catheter-associated urinary tract infection
Pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Headache/Delirium
Breathing Issues (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Shortness of breath
Closed displaced fracture of left tibial spine (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Immediate Start - Exercise Program (N=12) | Immediate Start - No Exercise (N=9) | Delayed Start - No Exercise (N=12) | Delayed Start - Exercise Program (N=8)
Pain (Musculoskeletal and connective tissue disorders) | 5 (13) | 0 (0) | 3 (3) | 5 (14)
Skin Issues (Skin and subcutaneous tissue disorders) | 4 (4) | 0 (0) | 0 (0) | 2 (4)
Breathing Issues (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sleep/mood disturbance (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infection (General disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Gastrointestinal Issues (Gastrointestinal disorders) | 1 (2) | 1 (1) | 0 (0) | 0 (0)
Lightheaded/Syncope (Ear and labyrinth disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Other (General disorders) | 1 (5) | 0 (0) | 0 (0) | 1 (2) — Falls, balance instability

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-08-14): https://cdn.clinicaltrials.gov/large-docs/49/NCT05376449/Prot_SAP_000.pdf